CLINICAL TRIAL: NCT00966316
Title: Establishment and Evaluation to the Effects of a Clinical Pathway for Acute Ischemic Stroke
Acronym: PAIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Yefeng,Cai, Guangdong Provincial Hospital of Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200707004
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke；clinical pathway;TCM；
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pathway (Experimental): aspirin，Chinese herbs；acupuncture；rehabilitation；health education；
  Interventions: Drug: aspirin，chinese herbs；

INTERVENTIONS:
Drug: aspirin，chinese herbs； — aspirin 300mg/100mg,qd,chinese herbs, one dose ，qd
  Other Names: Bayer

SUMMARY:
The purpose of this study is to determine whether the clinical pathway for acute ischemic stroke(with combination of traditional Chinese medicine and western medicine) is able to improve the outcome of acute ischemic stroke and evaluate its effect on hospital day and cost, etc. Meanwhile, the study will discuss the safety and efficiency of this kind of Clinical Pathway

DETAILED DESCRIPTION:
Eligibility Ages Eligible for Study: 18 Years to 85 Years Genders Eligible for Study: Both Accepts Healthy Volunteers: No

Criteria

Inclusion Criteria:

Those clinically diagnosed with acute ischemic stroke ； 18-85 years old； Over 6 hours and within 14 days from onset 4<=NIHSS <=22; Informed consent signed by patient or his/her family ；

Exclusion Criteria:

Hemorrhagic stroke; Cerebral hernia; Serious heart, liver, lung, kidney functional failure，malignancy; Not cooperative with physician; Psychological disorder; Already taken part in other clinical drug trial within the past 3 months

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke diagnosed with both criteria of traditional Chinese medicine and western medicine；
* 18-85 years old；
* Over 6 hours and within 14 days from onset
* 4<=NIHSS <=22;
* Informed consent signed by patient or his/her family ；

Exclusion Criteria:

* Hemorrhagic stroke;
* Cerebral hernia;
* Serious heart, liver, lung, kidney functional failure,malignancy;
* Not cooperative with physician;
* Psychological disorder;
* Already taken part in other clinical drug trial within the past 3 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
death rate；average hospital day；cost of hospitalization | 3 months；discharge day

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) National Institute of Health Stroke Scale (NIHSS) Barthel Index degree of satisfaction | 7 day；30 day；3 months

CONTACTS AND LOCATIONS:
Overall Officials: yefeng cai, postgraduate, Study Chair — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Adams HP Jr, del Zoppo G, Alberts MJ, Bhatt DL, Brass L, Furlan A, Grubb RL, Higashida RT, Jauch EC, Kidwell C, Lyden PD, Morgenstern LB, Qureshi AI, Rosenwasser RH, Scott PA, Wijdicks EF; American Heart Association/American Stroke Association Stroke Council; American Heart Association/American Stroke Association Clinical Cardiology Council; American Heart Association/American Stroke Association Cardiovascular Radiology and Intervention Council; Atherosclerotic Peripheral Vascular Disease Working Group; Quality of Care Outcomes in Research Interdisciplinary Working Group. Guidelines for the early management of adults with ischemic stroke: a guideline from the American Heart Association/American Stroke Association Stroke Council, Clinical Cardiology Council, Cardiovascular Radiology and Intervention Council, and the Atherosclerotic Peripheral Vascular Disease and Quality of Care Outcomes in Research Interdisciplinary Working Groups: The American Academy of Neurology affirms the value of this guideline as an educational tool for neurologists. Circulation. 2007 May 22;115(20):e478-534. doi: 10.1161/CIRCULATIONAHA.107.181486. PMID 17515473
- See also: Related Info — http://www.gdhtcm.com/